CLINICAL TRIAL: NCT00302471
Title: A Phase I, Randomized, Multicenter, Double-Blind Study of MK0429 in the Treatment of Men With Hormone Refractory Prostate Cancer and Metastatic Bone Disease
Brief Title: MK0429 Study in Prostate Cancer Patients With Metastatic Bone Disease (0429-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0429-011; MK0429-011; 2006_013
Record Dates: First submitted 2006-03-09; First posted 2006-03-14 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1600 mg twice a day (Experimental): MK0429
  Interventions: Drug: Comparator: MK0429
- 200 mg twice a day (Experimental): MK0429
  Interventions: Drug: Comparator: MK0429
- 800 mg twice a day (Experimental): MK0429
  Interventions: Drug: Comparator: MK0429
- 400 mg twice a day (Experimental): MK0429
  Interventions: Drug: Comparator: MK0429

INTERVENTIONS:
Drug: Comparator: MK0429 — Part 1 - MK3328 of 1600 mg twice a day for 4 weeks given to men with hormone refractory prostate cancer and metastatic bone.
  Disease.
  Arms: 1600 mg twice a day
Drug: Comparator: MK0429 — Part 2- MK3328 of 200 mg twice a day for 4 weeks to men with hormone refractory prostate cancer and metastatic bone disease.
  Arms: 200 mg twice a day
Drug: Comparator: MK0429 — Part 1- MK3328 of 800mg twice a day for 8 weeks to men with hormone refractory prostate cancer and metastatic bone disease.
  Arms: 800 mg twice a day
Drug: Comparator: MK0429 — Part 2 - MK3328 of 400 mg twice a day for 8 weeks to men with hormone refractory prostate cancer and metastatic bone disease.
  Arms: 400 mg twice a day

SUMMARY:
This two part study will evaluate the safety and tolerability of MK0429 in addition to assessing it's pharmacokinetic profile and pharmacodynamic response.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have:

  * Prostate cancer
  * Bone metastases without symptoms
  * Lack of response to hormone therapy as evidenced by a rising PSA or clinical progression

Exclusion Criteria:

* Prostate cancer-related bone pain
* Previously received bisphosphonate therapy (e.g. zoledronate)
* Received any investigational treatment within the last 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 4 weeks of MK0429 therapy. | up to 14 days following last dose of medication

SECONDARY OUTCOMES:
Part 1: Pharmacokinetic profile of MK0429 and pharmacodynamic responses to treatment of MK0429 | 4 weeks
Part 2: Pharmacokinetic profile of MK0429 [Time frame 4 weeks] and pharmacodynamic responses to treatment of MK0429 [Time frame 8 weeks] | 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Rosenthal MA, Davidson P, Rolland F, Campone M, Xue L, Han TH, Mehta A, Berd Y, He W, Lombardi A. Evaluation of the safety, pharmacokinetics and treatment effects of an alpha(nu)beta(3) integrin inhibitor on bone turnover and disease activity in men with hormone-refractory prostate cancer and bone metastases. Asia Pac J Clin Oncol. 2010 Mar;6(1):42-8. doi: 10.1111/j.1743-7563.2009.01266.x. PMID 20398037